CLINICAL TRIAL: NCT01862458
Title: Prospective Randomized Trial: Fibrinolysis With tPA (Tissue Plasminogen Activator) Versus tPA and DNAse in Children With Empyema
Brief Title: Empyema Treated With tPA & DNAse
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: funding difficulty
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Assoc Prof, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12120552; 12120552 (Other: Children's Mercy Hospital)
Record Dates: First submitted 2013-05-17; First posted 2013-05-24 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Empyema
Keywords: empyema; tPA; dornase
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tPA alone (Active Comparator): tPA alone used to treat empyema
  Interventions: Biological: tPA alone
- tPA plus dornase (Experimental): tPA plus dornase used to treat empyema
  Interventions: Biological: tPA plus dornase

INTERVENTIONS:
Biological: tPA alone
  Arms: tPA alone
Biological: tPA plus dornase
  Arms: tPA plus dornase

SUMMARY:
The objective of this study is to scientifically evaluate a new substrate for fibrinolysis compared to our standard tPA.

The hypothesis, driven by a recent prospective trial, is that tPA may benefit from the addition of DNAse.

The primary outcome variable between the two techniques will be length of hospitalization after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients less than 18 years of age requiring an intervention for empyema by one of the following:

* Septation or loculation seen on ultrasound or computed tomography or
* Greater than 10,000 white blood cells identified on pleural tap

Exclusion Criteria:

* Immunodeficiency process
* Secondary diagnosis or condition that will keep them in the hospital beyond the empyema
* Existing contraindications to chest tube
* Documented allergy to one of the study medications

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Length of stay | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States